CLINICAL TRIAL: NCT02804737
Title: Impact of Patient Education Website on the Quality of Outpatient Bowel Preparation for Colonoscopy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Enns, Principal Investigator, University of British Columbia
Other Study IDs: H14-00468
Record Dates: First submitted 2015-05-11; First posted 2016-06-17 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Web Group: Patients given web site (aiddly) instructions for colonoscopy
  Interventions: Device: Aiddly (Web Site)
- Paper Group: Patients given paper instructions for colonoscopy

INTERVENTIONS:
Device: Aiddly (Web Site) — A website designed to better educate patients on how to prepare for their colonoscopies
  Groups: Web Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the GI clinic's currently used web-based instructions at St. Paul's Hospital.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a relatively common and life threatening condition that affect one in thirteen individuals in their lifetime. Colonoscopy is the most used procedure to allow gastroenterologist to identify colorectal malignancies or precancerous lesions at an earlier stage, which affords a greater chance for cure. However, low bowel cleanliness hinders polyp detection rates and therefore colonoscopy effectiveness. In the past, the majority of the studies have focused on pharmacological factors to optimize bowel preparation quality. Recently, the non-pharmacological factors have been found to have significant increases in bowel preparation quality. The purpose of this study is to evaluate the effectiveness of the GI clinic's currently used web-based instructions at St. Paul's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a colonoscopy as outpatients

Exclusion Criteria:

* Unable to speak English
* Unwilling to participate in reading online materials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been scheduled for a colonoscopy as outpatients
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Web-based instructions | Time 0
  Determine the effectiveness of Web-based instructions patients in preparing for colonoscopy by comparing the percentage of patients that achieved an excellent Boston Bowel Preparation Score when following the web-based instructions compared to historical control of paper written instructions.

SECONDARY OUTCOMES:
Benefit of web-based instructions | Time 0
  Determine through a survey the benefit to patients of this method of education.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Rex DK. Dosing considerations in the use of sodium phosphate bowel preparations for colonoscopy. Ann Pharmacother. 2007 Sep;41(9):1466-75. doi: 10.1345/aph.1K206. Epub 2007 Jul 24. PMID 17652123
- [Background] Park JS, Sohn CI, Hwang SJ, Choi HS, Park JH, Kim HJ, Park DI, Cho YK, Jeon WK, Kim BI. Quality and effect of single dose versus split dose of polyethylene glycol bowel preparation for early-morning colonoscopy. Endoscopy. 2007 Jul;39(7):616-9. doi: 10.1055/s-2007-966434. PMID 17611916
- [Background] Unger RZ, Amstutz SP, Seo DH, Huffman M, Rex DK. Willingness to undergo split-dose bowel preparation for colonoscopy and compliance with split-dose instructions. Dig Dis Sci. 2010 Jul;55(7):2030-4. doi: 10.1007/s10620-009-1092-x. Epub 2010 Jan 16. PMID 20082216
- [Background] Winawer S, Fletcher R, Rex D, Bond J, Burt R, Ferrucci J, Ganiats T, Levin T, Woolf S, Johnson D, Kirk L, Litin S, Simmang C; Gastrointestinal Consortium Panel. Colorectal cancer screening and surveillance: clinical guidelines and rationale-Update based on new evidence. Gastroenterology. 2003 Feb;124(2):544-60. doi: 10.1053/gast.2003.50044. PMID 12557158
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Muller AD, Sonnenberg A. Protection by endoscopy against death from colorectal cancer. A case-control study among veterans. Arch Intern Med. 1995 Sep 11;155(16):1741-8. doi: 10.1001/archinte.1995.00430160065007. PMID 7654107
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Belsey J, Epstein O, Heresbach D. Systematic review: oral bowel preparation for colonoscopy. Aliment Pharmacol Ther. 2007 Feb 15;25(4):373-84. doi: 10.1111/j.1365-2036.2006.03212.x. PMID 17269992
- [Background] Tan JJ, Tjandra JJ. Which is the optimal bowel preparation for colonoscopy - a meta-analysis. Colorectal Dis. 2006 May;8(4):247-58. doi: 10.1111/j.1463-1318.2006.00970.x. PMID 16630226
- [Background] Holt EW, Yimam KK, Ma H, Shaw RE, Sundberg RA, Verhille MS. Patient tolerability of bowel preparation is associated with polyp detection rate during colonoscopy. J Gastrointestin Liver Dis. 2014 Jun;23(2):135-40. doi: 10.15403/jgld.2014.1121.232.ewh1. PMID 24949604
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Serper M, Gawron AJ, Smith SG, Pandit AA, Dahlke AR, Bojarski EA, Keswani RN, Wolf MS. Patient factors that affect quality of colonoscopy preparation. Clin Gastroenterol Hepatol. 2014 Mar;12(3):451-7. doi: 10.1016/j.cgh.2013.07.036. Epub 2013 Aug 15. PMID 23954647